CLINICAL TRIAL: NCT04092244
Title: CTHRC1 as a New Biomarker in Diagnosis of Rheumatoid Arthritis and Its Role in Seronegative Patients.
Brief Title: Role of CTHRC1 in Diagnosis of Rheumatoid Arthritis
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Amany Abdelkader Ahmed Hefny, Resident physician, Assiut University
Other Study IDs: CTHRC1 in rheumatoid disease
Record Dates: First submitted 2019-09-15; First posted 2019-09-17 (Actual); Last update posted 2020-05-28 (Actual); Status verified 2020-05

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: CTHRC1 biomarker — its a biomarker detected in the serum of the patients

SUMMARY:
to detect the role of CTHRC1 biomarker in diagnosis of rheumatoid arthritis and To correlate other well-established rheumatoid arthritis markers (RF& anti-ccp) and CTHRC1 level to see if CTHRC1 can act as a dependent or independent serum marker in prediction of RA status.

DETAILED DESCRIPTION:
Rheumatoid arthritis (RA) is a chronic, progressive, autoimmune disease of synovial joints. Disease progression is characterized by periods of high disease activity involving both, a systemic immune response and tissue-specific inflammatory events that may lead to joint and bone destruction and subsequent disability.

Rheumatoid arthritis is a multifactorial disease with significant contribution from genetic and non-genetic factors that together account for complex disease pathology.

Diagnosis of RA is based mainly on detection of high titers of rheumatoid factor (RF) and of antibodies against cyclic citrullinated peptide (anti-CCP) or against citrullinated protein (ACPA).

The major RF species could be detected only in 60-70% of RA patients; patients with high levels of RF have higher disease activity with greater disabilities.

The problem is that RF is not a specific marker for RA and is often absent in early stages of the disease, on the other hand ACPA and CCP auto antibodies provide high specificity but moderate sensitivity, adding to that CRP and ESR are general indicators of inflammation and are not specific for RA.

Collagen triple helix repeat containing 1 protein (CTHRC1) is expressed in a number of embryonic and neonate tissues, including developing cartilage and bone. It is a secreted modulator of Wnt signaling, which is a key regulator of joint remodeling and promotes cell proliferation and migration.

Immunohistochemical analysis of various human primary cancers and metastases has revealed that CTHRC1 expression is actually limited to the stromal cells of solid tumors.

The expression of CTHRC1 encoding gene was found to be strongly associated with the severity of murine collagen antibody-induced arthritis.

Arthritic pannus is a multicellular vascularized tissue composed of cells of both mesenchymal and hematopoietic origin, including synovial fibroblasts, osteoclasts, endothelial cells, dendritic cells, monocytes/macrophages, as well as T and B cells that contribute to the development and progression of joint and cartilage erosion through secretion of pro-inflammatory cytokines and tissue-degrading proteases. Fibroblast-like synoviocytes (FLS), particularly the invasive and migratory cadherin-11-positive subtype, are major components of synovial pannus tissue and are considered active drivers in the pathogenesis of RA.

The expression of CTHRC1 in pannus and its role in the function of FLS relevant to cartilage damage in RA make it of great value if used as a blood-based biomarker for improved diagnosis of rheumatoid arthritis patients.

ELIGIBILITY:
Inclusion Criteria:

* All RA patients must fulfill the 2010 ACR/EULAR criteria for RA.
* Healthy individual must be without a prior history of chronic inflammation or any form of arthritis.

Exclusion Criteria:

* - Patients with solid tumors.

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: The study will include the following:
  * 35 RA patients with negative anti_ccp.
  * 35 RA patients with negative RF.
  * 45 RA patients either positive RF or anti-ccp.
  * 30 other Arthritic patients.
  * 25 healthy controls.
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2020-08-01 (Estimated); Primary Completion 2021-11-28 (Estimated); Study Completion 2021-12-30 (Estimated)

PRIMARY OUTCOMES:
detect value of CTHRC1 in diagnosis of rheumatoid arthritis | baseline
  detect the role of CTHRC1 biomarker in diagnosis of rheumatoid arthritis and To compare the sensitivity and the specificity of CTHRC1 in relation to other biomarkers used in diagnosis of RA.

REFERENCES:
- [Background] Smolen JS, Aletaha D, Barton A, Burmester GR, Emery P, Firestein GS, Kavanaugh A, McInnes IB, Solomon DH, Strand V, Yamamoto K. Rheumatoid arthritis. Nat Rev Dis Primers. 2018 Feb 8;4:18001. doi: 10.1038/nrdp.2018.1. PMID 29417936
- [Background] Shekhani MT, Forde TS, Adilbayeva A, Ramez M, Myngbay A, Bexeitov Y, Lindner V, Adarichev VA. Collagen triple helix repeat containing 1 is a new promigratory marker of arthritic pannus. Arthritis Res Ther. 2016 Jul 19;18:171. doi: 10.1186/s13075-016-1067-1. PMID 27430622
- [Background] Song YW, Kang EH. Autoantibodies in rheumatoid arthritis: rheumatoid factors and anticitrullinated protein antibodies. QJM. 2010 Mar;103(3):139-46. doi: 10.1093/qjmed/hcp165. Epub 2009 Nov 19. PMID 19926660
- [Background] Singal DP, Li J, Zhu Y. Genetic basis for rheumatoid arthritis. Arch Immunol Ther Exp (Warsz). 1999;47(5):307-11. PMID 10604236
- [Background] Nell VP, Machold KP, Stamm TA, Eberl G, Heinzl H, Uffmann M, Smolen JS, Steiner G. Autoantibody profiling as early diagnostic and prognostic tool for rheumatoid arthritis. Ann Rheum Dis. 2005 Dec;64(12):1731-6. doi: 10.1136/ard.2005.035691. Epub 2005 May 5. PMID 15878904
- [Background] Lefevre S, Knedla A, Tennie C, Kampmann A, Wunrau C, Dinser R, Korb A, Schnaker EM, Tarner IH, Robbins PD, Evans CH, Sturz H, Steinmeyer J, Gay S, Scholmerich J, Pap T, Muller-Ladner U, Neumann E. Synovial fibroblasts spread rheumatoid arthritis to unaffected joints. Nat Med. 2009 Dec;15(12):1414-20. doi: 10.1038/nm.2050. Epub 2009 Nov 8. PMID 19898488
- [Background] Han B, Pouget JG, Slowikowski K, Stahl E, Lee CH, Diogo D, Hu X, Park YR, Kim E, Gregersen PK, Dahlqvist SR, Worthington J, Martin J, Eyre S, Klareskog L, Huizinga T, Chen WM, Onengut-Gumuscu S, Rich SS; Major Depressive Disorder Working Group of the Psychiatric Genomics Consortium; Wray NR, Raychaudhuri S. A method to decipher pleiotropy by detecting underlying heterogeneity driven by hidden subgroups applied to autoimmune and neuropsychiatric diseases. Nat Genet. 2016 Jul;48(7):803-10. doi: 10.1038/ng.3572. Epub 2016 May 16. PMID 27182969
- [Background] Durmus T, LeClair RJ, Park KS, Terzic A, Yoon JK, Lindner V. Expression analysis of the novel gene collagen triple helix repeat containing-1 (Cthrc1). Gene Expr Patterns. 2006 Oct;6(8):935-40. doi: 10.1016/j.modgep.2006.03.008. Epub 2006 Mar 17. PMID 16678498
- [Background] Ding B, Padyukov L, Lundstrom E, Seielstad M, Plenge RM, Oksenberg JR, Gregersen PK, Alfredsson L, Klareskog L. Different patterns of associations with anti-citrullinated protein antibody-positive and anti-citrullinated protein antibody-negative rheumatoid arthritis in the extended major histocompatibility complex region. Arthritis Rheum. 2009 Jan;60(1):30-8. doi: 10.1002/art.24135. PMID 19116921